CLINICAL TRIAL: NCT03145467
Title: Comparison of Oral Paracetamol and Zolmitriptan Efficacy in the Treatment of Acute Migraine Headache in Emergency Department: Randomize Controlled Trial
Brief Title: Comparison of Oral Paracetamol and Zolmitriptan Efficacy in the Treatment of Acute Migraine in Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ibrahim Turkcuer, professor, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015TPF039
Record Dates: First submitted 2017-04-21; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acute Migraine Headache
Keywords: Migraine; Paracetamol; Zolmitriptan; Emergency services
MeSH Terms: conditions — Migraine Disorders | interventions — Acetaminophen; zolmitriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol (Experimental): 1000 mg of paracetamol (Parol Tablet - Atabay İlaç Fabrikası A.Ş.) Oral (PO) was given 100 patients
  Interventions: Drug: Paracetamol
- Zolmitriptan (Experimental): Second Group: Zolmitirptan 2,5 mg (Zomig Tablet - Astra Zeneca) oral (PO) was given 100 patients.
  Interventions: Drug: Zolmitriptan

INTERVENTIONS:
Drug: Paracetamol — 1000 mg of paracetamol (Parol Tablet - Atabay İlaç Fabrikası A.Ş.) Oral (PO) was given 100 patients
  Other Names: Parol
  Arms: Paracetamol
Drug: Zolmitriptan — Zolmitirptan 2,5 mg (Zomig Tablet - Astra Zeneca) oral (PO) was given 100 patients
  Other Names: Zomig
  Arms: Zolmitriptan

SUMMARY:
Migraine is a chronic and sometimes progressive disorder, characterized by headache, recurrent episodes, and other associated symptoms. Migraine is the most common cause of headache among patients who applied to emergency services.

The purpose of the investigators is to compare the efficacy of oral paracetamol and zolmitriptan in the treatment of acute migraine headache in an emergency department.

DETAILED DESCRIPTION:
* This is prospective, randomized, controlled research to compare the efficacy of these two drugs in emergancy department.
* The clinical trial was conducted in the ED of Pamukkale University Medical Faculty Hospital.
* Study personnel (emergency physicians and nurses) were trained before the study.
* When oral drugs (paracetamol, zolmitriptan was being recommended, an eligibility checklist was completed by the attending physician.
* If there were no exclusion criteria, written informed consent was obtained and baseline information, including initial headache pain score ratings with VAS and NRS were recorded.
* The need for identification and enrollment of participants by staff with conflicting work pressures resulted in recruitment of a convenience sample of patients.
* All patients eligible for the study were randomized to one of two groups:
* First Group: paracetamol 1000 mg was given oral to 100 patients,
* Second Group: Zolmitriptan 2,5 mg was given oral to 100 patients which determined to be applied as a group.
* Drugs were prepared according to the computer-generated random number sequence to assign treatment allocations.
* The allocation list was kept by the emergency nurse. Patients received the paracetamol, zolmitriptan medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug was obtained, and administered as oral.
* Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms)
* One researcher blinded to patient allocation observed the whole procedure and recorded the Headache scores.
* Headache scores were recorded at 0, 15, 30, and 60 min on a VAS of 1 to 100 mm and NRS of 1 to 10. Patients with nausea are treated with 15 minutes of 10 mg metoclorpramide slow infusion in 150 cc saline solution.
* Rescue medication (1 mcg/kg fentanyl ) was given İntravenöz to patients if pain VAS scores ≥ 50 mm in 60 minutes after study drug administration.
* All other medications required during the study also were recorded.
* During the study, pulse rate, systolic blood pressure, diastolic blood pressure, respiration rate and oxygen saturation (SpO2) were recorded at baseline (0 min), 15, 30, and 60 min.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were aged 18 years or older, 65 years or younger
* Had acute migraine attack without aura
* VAS (visual analog scale) score >50 mm , NRS (Numeric Rating Scale) score >5
* Patients whose written consent is obtained by agreeing to participate in the study

Exclusion Criteria:

* Those who refuse to participate in the work
* Patients younger than 18 years or older than 65 years
* Those who use ergotamine derivative drugs in the last 24 hours
* Have received analgesics in the last 6 hours
* Patients with severe liver, kidney, lung and heart failure
* To have active peptic ulcer bleeding or perforation
* Have a history of upper gastrointestinal disease
* To be Pregnancy and breast-feeding
* Patients of childbearing age who are not using a birth control method.
* Allergy to medicines used in work
* Hemodynamically unstable patients
* Patients with renal transplantation
* Blood pressure uncontrolled hypertension patients
* Patients with cerebrovascular disease history
* Patients with ischemic heart disease or coronary spasm / printzmetal angina
* Patients with arrhythmia accompanying Wolff-Parkinson-White syndrome or accessory conduits in the heart
* Patients with Glucose 6 Phosphate Dehydrogenase (G6PD) deficiency
* Those with other systemic diseases,
* Patients with a Visual Analogue Scale (VAS) pain score less than 50 mm
* Illiterates and patients with vision problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Decrement of the pain on VAS | Change from baseline in migraine headache VAS score at 60 minutes
  1. Compare decrease of migraine headache VAS (visual analog scale) score between the two groups. - (First group Paracetamol and Second Zolmitriptan)
Decrement of the pain on NRS | Change from baseline in migraine headache NRS score at 60 minutes
  1. Compare decrease of migraine headache NRS (Numeric Rating Scale) score between the two groups. - (First group Paracetamol and Second Zolmitriptan)

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt Arikan, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No